CLINICAL TRIAL: NCT01599234
Title: A Double Blind, Randomised, Placebo Controlled, Parallel Group Study of Sativex, in Subjects With Symptoms of Spasticity Due to Multiple Sclerosis.
Brief Title: A Study to Evaluate the Efficacy of Sativex in Relieving Symptoms of Spasticity Due to Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWCL0403
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental): Active treatment
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — Contains delta-9-tetrahydrocannabinol (THC) (27mg/ml): cannabidiol (CBD) (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg:CBD 60 mg) in 24 hours.
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — Contains peppermint oil flavouring, 0.05%(v/v); quinoline yellow,0.005% (w/v) and sunset yellow, 0.0025% (w/v) colourants, in a and ethanol:propylene glycol (50:50) excipient.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the efficacy of Sativex in relieving symptoms of spasticity in multiple sclerosis

DETAILED DESCRIPTION:
This was a 15 week (one week baseline and fourteen weeks treatment period), multicentre, double blind, randomised, placebo controlled, parallel group study to evaluate the efficacy of Sativex in subjects with symptoms of spasticity due to multiple sclerosis. Eligible subjects entered a seven day baseline period. Subjects then returned to the centre for randomisation and dose introduction. Visits occurred at the end of treatment weeks two, six, ten and at the end of the study (treatment week 14) or earlier if they withdrew.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Aged 18 years or above.
* Ability (in the investigator's opinion) and willingness to comply with all study requirements.
* Diagnosed with any disease subtype of multiple sclerosis of duration greater than six months.
* Diagnosed with spasticity due to multiple sclerosis of at least three months duration and was not wholly relieved with their current therapy.
* Stable dose of anti-spasticity and non-pharmacological therapies for at least 30 days prior to the screening visit and willingness for these to be maintained for the duration of the study.
* Stable dose of disease modifying medications for at least six months duration prior to the screening visit and willingness to maintain this for the duration of the study.
* The last six daily diary spasticity numerical rating scale scores before randomisation had been completed and summed to at least 24.
* Agreement for the responsible authorities (as applicable in individual countries), their primary care physician, and their consultant, if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* Concomitant disease or disorder that had symptoms of spasticity, or that may have influenced the subject's level of spasticity.
* Received a Botulinum Toxin injection within four months prior to the screening visit or unwillingness to stop receiving Botulinum Toxin injections for the relief of spasticity for the duration of the study.
* Had used cannabis within 30 days of study entry and unwillingness to abstain for the duration for the study.
* Had used cannabinoid based medications within 60 days of study entry and unwillingness to abstain for the duration for the study.
* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Known or suspected history of alcohol or substance abuse.
* History of epilepsy or recurrent seizures.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medication.
* Experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction.
* QT interval of > 450 ms (males) or > 470 ms (females) at Visit 1.
* Secondary to tertiary arterial ventricular block or sinus bradycardia (heart rate < 50 bpm) or sinus tachycardia (heart rate > 110 bpm) at Visit 1.
* Diastolic blood pressure of < 50 mmHg or > 105 mmHg in a sitting position at rest for 5 minutes prior to randomisation.
* Impaired renal function i.e. serum creatinine clearance is lower than 50 ml/min at Visit 1.
* Significantly impaired hepatic function, at Visit 1, in the investigator's opinion and/or had liver function tests of equal to or greater than three times the upper limit of normal.
* Female subjects of child bearing potential and male subjects whose partner was of child bearing potential, unless were willing to ensure that they or their partner used effective contraception during the study and for three months thereafter.
* If female, were pregnant or lactating, or were planning pregnancy during the course of the study and for three months thereafter.
* Received an IMP within the 12 weeks before Visit 1.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical examination, the subject had any abnormalities that, in the opinion of the investigator, would prevent the subject from safely participating in the study.
* Scheduled elective surgery or other procedures, which required general anaesthesia during the study.
* Intention to donate blood during the study.
* Intention to travel internationally during the study.
* Previous randomisation into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Collin, Principal Investigator — The Royal Berkshire and Battle Hospitals NHS Trust, London Road, Reading, Berkshire, RG1 5AN.
Locations (1):
- The Royal Berkshire and Battle Hospitals NHS Trust, Reading, United Kingdom

REFERENCES:
- [Result] Collin C, Ehler E, Waberzinek G, Alsindi Z, Davies P, Powell K, Notcutt W, O'Leary C, Ratcliffe S, Novakova I, Zapletalova O, Pikova J, Ambler Z. A double-blind, randomized, placebo-controlled, parallel-group study of Sativex, in subjects with symptoms of spasticity due to multiple sclerosis. Neurol Res. 2010 Jun;32(5):451-9. doi: 10.1179/016164109X12590518685660. Epub 2010 Mar 19. PMID 20307378
- [Derived] Di Marzo V, Centonze D. Placebo effects in a multiple sclerosis spasticity enriched clinical trial with the oromucosal cannabinoid spray (THC/CBD): dimension and possible causes. CNS Neurosci Ther. 2015 Mar;21(3):215-21. doi: 10.1111/cns.12358. Epub 2014 Dec 4. PMID 25475413

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours.
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 24 actuations in 24 hours.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 167 | 170
Completed | 150 | 155
Not Completed | 17 | 15
Not completed — Adverse Event | 9 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 2 | 4
Not completed — Unable to operate spray | 1 | 0
Not completed — Sponsor request as creatinine levels <50 | 0 | 1
Not completed — Death | 1 | 0
Not completed — Patient would not stop driving | 1 | 0
Not completed — Contra-indication discovered | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 167 | 170 | 337
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 162 | 168 | 330
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (10.06) | 47.1 (9.15) | 47.5 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 101 | 207
  Male | 61 | 69 | 130
Region of Enrollment [Number; unit: participants]
  United Kingdom | 65 | 63 | 128
  Czech Republic | 102 | 107 | 209

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Spasticity 0-10 Numerical Rating Scale (NRS) Score During the Last 14 Day of Treatment (End of Treatment)
Description: The average spasticity NRS was completed at the same time each day, i.e. bedtime in the evening. The subject was asked "on a scale of '0 to 10', please indicate the number that best describes your spasticity in the last 24 hours" where 0 = no spasticity and 10 = worst possible spasticity. A negative value indicates an improvement in pain score from baseline.
Time Frame: 0-15 weeks
Population: All subjects who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 166 | 169
units on a scale | -1.22 (1.76) | -0.91 (1.72)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The initial model used for the analysis of the end of study value was an analysis of covariance (ANCOVA) with baseline as a covariate and treatment group, centre group, ambulatory status at baseline and previous use of cannabis as main effects. Interactions between the main effects were investigated, and if they had little influence then they were dropped from the model. These tests were performed at the 10% significance level as a possible indicator of an interactive effect; Test type: Superiority or Other; p = 0.220, ANCOVA; Estimated mean treatment difference = -0.23, 95% CI [-0.59 to 0.14]

2. Secondary Outcome: Number of Subjects With a 30% or Greater Improvement in Mean Spasticity 0-10 NRS Score at the End of Treatment Compared to Baseline
Description: The cumulative response to treatment was the percentage change from baseline in the mean NRS spasticity score as defined as the 30% response. The spasticity NRS was completed at the same time each day, i.e. bedtime in the evening. The subject was asked "on a scale of '0 to 10', please indicate the number that best describes your spasticity in the last 24 hours" where 0 = no spasticity and 10 = worst possible spasticity. The number of responders at the 30% level is presented.
Time Frame: 0-15 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 166 | 169
participants | 51 | 42
Statistical Analysis 1: Comparison: Sativex vs Placebo; The numbers of responders was analysed using the difference in proportions and the odds ratio comparing the treatment groups with the provision of 95% CIs for the difference and odds ratio. The two groups were compared using ANCOVA with baseline severity as a covariate and study centre and treatment group as factors; Test type: Superiority or Other; p = 0.231, ANCOVA; Odds Ratio (OR) = 1.341, 95% CI 2-sided [0.830 to 2.167]

3. Secondary Outcome: Change From Baseline in the Mean Modified Ashworth Scale Score at the End of Treatment
Description: All 20 muscle groups were assessed for spasticity (using a 1-5 scale): 1= no increase in muscle tone to 5= passive movement is difficult and affected part is rigid in flexion or extension. The score for all 20 muscle groups were added to give a total score out of 100; minimum score was 20. A decrease in score indicates an improvement in condition.
Time Frame: Day 0 (Randomisation) and Day 99 (End of Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 156 | 160
units on a scale | -3.3 (9.25) | -2.8 (7.81)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment, centre group and ambulatory status at baseline as factors and baseline score as a covariate; Test type: Superiority or Other; p = 0.857, ANCOVA; Estimated mean treatment difference = -0.16, 95% CI 2-sided [-1.94 to 1.61]

4. Secondary Outcome: Change From Baseline in Mean Sleep Quality 0-10 NRS During the Last 14 Days of Treatment (End of Treatment)
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The subject was asked "on a scale of '0 to 10', please indicate how your spasticity disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: 0-15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 124 | 139
units on a scale | -0.7 (2.85) | -0.6 (2.37)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The two groups were compared using ANCOVA with baseline severity as a covariate and study centre and treatment group as factors; Test type: Superiority or Other; p = 0.734, ANCOVA; Estimated mean treatment difference = -0.07, 95% CI 2-sided [-0.55 to 0.40]

5. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who experienced and adverse event during the course of the study is presented
Time Frame: 0-15 weeks
Population: All subjects who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the analysis, as were a further two subjects who were excluded from the full analysis set (used for the efficacy analysis) as a result of no on-treatment efficacy data
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 170
participants | 156 | 132

6. Secondary Outcome: Change From Baseline in Mean Timed 10 Metre Walk Time at the End of Treatment
Description: Only those subjects for whom it was appropriate (i.e. ambulatory subjects) were timed how long it took to walk 10 metres. Walk time was only assessed for subjects who successfully completed the Timed 10 Metre Walk. A negative difference from baseline indicates an improvement walk time.
Time Frame: Day 0 (Randomisation) and Day 99 (End of Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 115 | 120
time (seconds) | -2.1 (17.37) | 9.3 (63.56)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change at end of treatment was compared between treatment groups using ANCOVA. The model included treatment, centre group and ambulatory status at baseline as factors and baseline score as a covariate; Test type: Superiority or Other; p = 0.624, ANCOVA; Estimated mean treatment difference = 0.0, 95% CI 2-sided [-2.0 to 1.0]

7. Secondary Outcome: Carer Global Impression of Change at the End of Treatment
Description: The carer of the subject gave their opinion of any noticeable change in the subject's overall functional ability at the end of the study. A 7-point Likert-type scale was used, with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". The number of carers who reported an improvement at the end of treatment is presented.
Time Frame: Day 99 (end of treatment)
Population: All subjects who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the analysis, as were a further two subjects who were excluded from the full analysis set as a result of no on-treatment efficacy data
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 170
participants | 72 | 56
Statistical Analysis 1: Comparison: Sativex vs Placebo; The two treatment groups were to be compared using ordinal logistic regression and the proportional odds model. The model was to incorporate ambulatory status at baseline and centre group; Test type: Superiority or Other; p = 0.270, Regression, Logistic; Odds Ratio (OR) = 1.248, 95% CI 2-sided [0.842 to 1.849]

8. Secondary Outcome: Change From Baseline in the Mean Total Barthel Activities of Daily Living Index Score at the End of Treatment
Description: The Barthel Index consists of 10 items that measure a person's daily functioning specifically the activities of daily living and mobility. The items include feeding, moving from wheelchair to bed and return, grooming, transferring to and from a toilet, bathing, walking on level surface, going up and down stairs, dressing, continence of bowels and bladder. The person receives a score based on whether they have received help while doing the task. The scores for each of the items are summed to create a total score of 100. An increase in score indicates an improvement.
Time Frame: Day 0 (Randomisation) and Day 99 (End of Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 162 | 165
units on a scale | -0.1 (10.26) | 0.5 (8.05)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.867, ANCOVA; Estimated mean treatment difference = -0.15, 95% CI 2-sided [-1.95 to 1.64]

9. Secondary Outcome: Number of Subjects With a 50% or Greater Improvement in Mean Spasticity 0-10 NRS Score at the End of Treatment Compared to Baseline
Description: The cumulative response to treatment was the percentage change from baseline in the mean NRS spasticity score as defined as the 50% response. The spasticity NRS was completed at the same time each day, i.e. bedtime in the evening. The subject was asked "on a scale of '0 to 10', please indicate the number that best describes your spasticity in the last 24 hours" where 0 = no spasticity and 10 = worst possible spasticity. The number of responders at the 50% level is presented.
Time Frame: 0 - 15 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 166 | 169
participants | 21 | 18
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.569, ANCOVA; Odds Ratio (OR) = 1.215, 95% CI 2-sided [0.622 to 2.373]

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up were collected (Days 0 - 134). All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 15/167 | 7/170
Other Adverse Events (participants affected / at risk) | 156/167 | 132/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=167) | Placebo (N=170)
Irritability (General disorders) | 1 | 0 — Irritability may have been misclassified to the General Disorders and Administration Site Conditions SOC from the Psychiatric Disorders SOC.
Asthenia (General disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 2
Orchitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 2
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Muscle Spasticity (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Drug Dependence (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Delusions (Psychiatric disorders) | 1 | 0
Depression Worsened (Psychiatric disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Phlebothrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=167) | Placebo (N=170)
Dizziness (Nervous system disorders) | 53 | 17
Somnolence (Nervous system disorders) | 24 | 7
Muscle Spasticity (Nervous system disorders) | 17 | 13
Headache (Nervous system disorders) | 15 | 10
Dysgeusia (Nervous system disorders) | 9 | 0
Disturbance in Attention (Nervous system disorders) | 7 | 0
Dysarthria (Nervous system disorders) | 7 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 5 | 5
Fatigue (General disorders) | 42 | 32
Asthenia (General disorders) | 26 | 11
Feeling Abnormal (General disorders) | 6 | 1
Malaise (General disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 53 | 17
Dry Mouth (Gastrointestinal disorders) | 24 | 7
Diarrhoea (Gastrointestinal disorders) | 15 | 10
Vomiting (Gastrointestinal disorders) | 9 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 7 | 0
Insomnia (Psychiatric disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 5
Urinary Tract Infection Not Otherwise Specified (Infections and infestations) | 19 | 21
Vertigo (Ear and labyrinth disorders) | 19 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.